CLINICAL TRIAL: NCT01257321
Title: Risk Stratification of Post Tonsillectomy Respiratory Complications in the Pediatric Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: OSA-HMO-CTIL
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Post Tonsillectomy Respiratory Complications

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (1):
- post tonsillectomy: children

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is the most common indication for tonsillectomy and adenoidectomy in young children. According to previous studies, as much as 8 to 20% of patients will develop post operative respiratory complications requiring medical intervention. The pre-operative risk factors that could predict respiratory complications retrospectively analyzed were young age, obesity and high preoperative apnea-hypopnea index. Despite the removal of obstructing lymphoid tissue, upper airway obstruction occurs on the first postoperative night in children with OSA. There is a debate regarding the post-operative duration and monitoring needed in children with OSA.

Hypothesis:

Pre-operative, operative and immediate post-operative parameters could predict post tonsillectomy respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patient < 14 years old
2. Obstructive sleep apnea according to polysomnography
3. Surgery: Tonsillectomy/Tonsillotomy

Exclusion Criteria:

1. Patient suffering from known respiratory disease

Max Age: 14 Years | Sex: All
Age Groups: Child
Study Population: children, suffering of obstructive sleep apnea, having their tonsills removed
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
respiratory distress

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel